CLINICAL TRIAL: NCT05658211
Title: Culture Analysis Performed During a Latarjet Anterior Shoulder Stabilization Procedure.
Acronym: CISAL
Status: Completed | Type: Observational
Sponsor: GCS Ramsay Santé pour l'Enseignement et la Recherche (Other)
Responsible Party: Sponsor
Other Study IDs: COS-RGDS-2021-06-014
Record Dates: First submitted 2022-11-25; First posted 2022-12-20 (Actual); Last update posted 2022-12-20 (Actual); Status verified 2022-11

CONDITIONS: Shoulder Instability Subluxation Bilateral

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a multicenter study of data from the medical records of patients who underwent shoulder stabilization surgery and who underwent a normally scheduled evaluation as part of their postoperative follow-up six months after surgery.

DETAILED DESCRIPTION:
Infection is a major cause of failure in shoulder arthroplasty and must be systematically sought at the time of revision, even if this is motivated by other complications (loosening, instability, periprosthetic fracture).

These cultures, performed in patients without clinical suspicion of infection, reveal, in 25 to 60% of cases, the presence of germs of cutaneous origin which, although generally considered to be non-virulent, continue to be debated as to their clinical significance and their implication in the failure of shoulder arthroplasty. Among these germs, propionibacterium acnes, staphylococcus epidermidis or coagulasenegative Staphylococcus are the most frequently identified.

The origin of these germs is still debated. Cultures of deep synovial fluid or tissues from patients receiving a first-line shoulder prosthesis show the presence of Cutibacterium acnes in 9% to 41% of cases despite preoperative antibiotic prophylaxis. These infections could be the consequence of contamination by a commensal germ during surgical exposure. Other authors consider them as an etiological factor in the development of shoulder arthritis. They would be more frequent in young subjects and male subjects.

The Latarjet procedure or coracoid bone block is commonly used in the surgical treatment of anterior shoulder instability.

It consists of cutting the coracoid bone with the coraco-biceps muscle that inserts on it, then passing it through the subscapularis muscle and fixing it on the scapula, thus creating a bone block. It can be performed by a conventional mini-invasive technique after an incision of 4 to 5 cm on the front of the shoulder or by arthroscopy.

The Latarjet procedure or coracoid bone block is commonly used in the surgical treatment of anterior shoulder instability.

It consists of cutting the coracoid bone with the coraco-biceps muscle that inserts on it, then passing it through the subscapularis muscle and fixing it on the scapula, thus creating a bone block. It can be performed by a conventional mini-invasive technique after an incision of 4 to 5 cm on the front of the shoulder or by arthroscopy.

ELIGIBILITY:
Inclusion Criteria:

* Patient 18 years of age or older, who has been informed of the research
* Patient who has undergone a first-line Latarjet operation
* Patient with three cultures performed on the coracoid bone blocks
* Patient regularly followed since the operation and for whom all data are available during the six-month follow-up visit.

Exclusion Criteria:

* Previous open shoulder surgery
* Associated rotator cuff injury requiring repair
* Clinical signs of preoperative infection
* Patient under court protection, guardianship or curatorship
* Patient who has indicated his or her opposition to the use of his or her medical data (by filling out and returning the non-opposition form that will be sent to him or her).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with no history of previous shoulder surgery or suspicion of underlying infection, operated on in the first instance for anterior shoulder instability by the conventional Latarjet technique (open surgery).
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2022-11-30 (Actual)

PRIMARY OUTCOMES:
Number of patients with positive culture | Month 6
  The primary endpoint, based on the culture result, is the number of patients with at least one positive culture

SECONDARY OUTCOMES:
Walch-Duplay Questionnaire | Month 6
  The Walch questionnaire includes a descriptive part (type and level of sport practiced, dominant score) and an evaluation scale of subjective and objective data (stability, pain, recovery of sport level, mobility) to assess the clinical result of the shoulder stabilization. The score ranges from 0 to 100. The result is considered excellent for a score of 91 to 100 points, good for 76 to 90 points, average for 51 to 75 points, and poor for a score of 50 points or less.
Constant score | Month 6
  The Constant and Murley score explores several domains: pain, activity, strength and mobility.
  The total score varies from 0 to 100 points, 100 points corresponding to a normal shoulder and 0 to a totally deficient shoulder.
Bacteriological criterion | Month 6
  Nature of germs identified in culture

CONTACTS AND LOCATIONS:
Locations (1):
- Clinique du Sport, Paris, France

IPD SHARING:
Plan to Share IPD: No